CLINICAL TRIAL: NCT00412217
Title: Phase III Randomized, Controlled Trial of Erlotinib (Tarceva) as Maintenance Therapy in Patients With Squamous Cell Carcinoma of the Head and Neck Treated With Resection and Radiotherapy With or Without Concomitant Chemotherapy With Curative Aim
Brief Title: A Study of Erlotinib (Tarceva) in Participants With Resected Head and Neck Squamous Cell Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated because recruitment was too slow.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML20294; 2006-001845-33 (EudraCT Number)
Record Dates: First submitted 2006-12-15; First posted 2006-12-18 (Estimated); Results first posted 2016-09-26 (Estimated); Last update posted 2016-11-25 (Estimated); Status verified 2016-10

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Erlotinib Hydrochloride; Standard of Care

ARMS (2):
- Erlotinib (Experimental): Participants treated with surgical resection and chemoradiotherapy or radiotherapy alone will receive erlotinib tablets as 150 mg PO daily for 1 year until disease progression or intolerable toxicity.
  Interventions: Drug: Erlotinib; Other: Standard of care
- Placebo (Placebo Comparator): Participants treated with surgical resection and chemoradiotherapy or radiotherapy alone will receive placebo treatment for 1 year until disease progression or intolerable toxicity.
  Interventions: Drug: Placebo; Other: Standard of care

INTERVENTIONS:
Drug: Placebo — Participants will receive placebo tablets (matched to erlotinib) once daily.
  Arms: Placebo
Drug: Erlotinib — Erlotinib will be given as 150 mg PO once daily.
  Other Names: Tarceva
  Arms: Erlotinib
Other: Standard of care — Additional clinical management including surgical resection and chemoradiotherapy or radiotherapy alone will be at the discretion of the Investigator according to local standard of care.

SUMMARY:
This two-arm study will compare the efficacy and safety of erlotinib (Tarceva) versus placebo in participants with resected head and neck squamous cell cancer who are receiving concurrent chemoradiotherapy or radiotherapy alone. Participants will be randomized to receive either erlotinib 150 milligrams (mg) orally (PO) once daily or placebo for 1 year until disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Adults greater than or equal to (≥) 18 years of age
* Curatively treated head and neck squamous cell cancer with T3-T4 and/or N2-N3 pathology, with or without other findings of poor prognosis such as extranodal extension, positive resection margins, and perineural or vascular involvement
* Eastern Cooperative Oncology Group (ECOG) status of 0 to 2

Exclusion Criteria:

* Macroscopic residual disease after surgery
* Previous treatment with anti-epidermal growth factor receptor (anti-EGFR) targeted therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2006-11; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (20):
- Spain (20):
  - Alcorcón
  - Barcelona
  - Burgos
  - Córdoba
  - Donostia / San Sebastian
  - Granada
  - Guadalajara
  - Jaén
  - Lugo
  - Madrid
  - Murcia
  - Ourense
  - Palma de Mallorca
  - Salamanca
  - Santander
  - Seville
  - Toledo
  - Valencia
  - Zamora
  - Zaragoza

RESULTS

PARTICIPANT FLOW:
Groups:
- Erlotinib: Participants with histologically confirmed advanced squamous cell carcinoma (SCC) of the head and neck, treated with surgical resection and chemoradiotherapy or radiotherapy alone, received erlotinib tablets as 150 milligrams (mg) once daily for 1 year until disease progression or intolerable toxicity.
- Placebo: Participants with histologically confirmed advanced SCC of the head and neck, treated with surgical resection and chemoradiotherapy or radiotherapy alone, received placebo tablets (matched to erlotinib) once daily for 1 year until disease progression or intolerable toxicity.
Period: Overall Study
Arm/Group | Erlotinib | Placebo
Started | 46 | 48
Completed | 0 | 0
Not Completed | 46 | 48
Not completed — Insufficient Data Available | 8 | 3
Not completed — Death | 5 | 4
Not completed — Disease Progression | 2 | 3
Not completed — Investigator Decision | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Lost to Follow-up | 1 | 4
Not completed — Study Terminated by Sponsor | 26 | 33
Not completed — Other | 1 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Population: All participants who were randomized in the study.
Groups:
- Erlotinib: Participants with histologically confirmed advanced SCC of the head and neck, treated with surgical resection and chemoradiotherapy or radiotherapy alone, received erlotinib tablets as 150 mg once daily for 1 year until disease progression or intolerable toxicity.
- Total: Total of all reporting groups
Arm/Group | Erlotinib | Placebo | Total
Number analyzed (Participants) | 46 | 48 | 94
Age, Customized [Number; unit: participants]
  18 Years or Older | 46 | 48 | 94
Sex/Gender, Customized [Number; unit: participants]
  Female | 3 | 7 | 10
  Male | 42 | 41 | 83
  Unknown | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Disease Progression
Description: Tumor response was assessed by the Investigator according to standard-of-care criteria, as there were no protocol-specified criteria for the assessment of tumor response and the instrument for assessment was deferred to the Investigator. To ensure comparability, baseline radiological studies later used to verify progression must be performed using identical techniques. The number of participants who experienced disease progression was reported.
Time Frame: From inclusion in the study until disease progression (maximum up to 3 years overall)
Population: ITT Population.
Measure: Number; unit: participants
Arm/Group | Erlotinib | Placebo
Number analyzed (Participants) | 46 | 48
participants | 15 | 11

2. Primary Outcome: Time to Progression (TTP)
Description: Tumor response was assessed by the Investigator according to standard-of-care criteria, as there were no protocol-specified criteria for the assessment of tumor response and the instrument for assessment was deferred to the Investigator. TTP was defined as the time from inclusion in the study to the time of disease progression, appearance of second tumor, or death from any cause, whichever occurred first. To ensure comparability, baseline radiological studies later used to verify progression must be performed using identical techniques. The median duration of TTP and corresponding 95% confidence interval (CI) were to be estimated by Kaplan-Meier analysis and expressed in months.
Time Frame: From inclusion in the study until disease progression, appearance of second tumor, or death from any cause (maximum up to 3 years overall)
Population: ITT Population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Erlotinib | Placebo
Number analyzed (Participants) | 46 | 48
months | NA [13.6259 to NA] — The median and upper limit of the 95% CI for PFS were not reached during the study period and could not be calculated. | NA [18.4110 to NA] — The median and upper limit of the 95% CI for PFS were not reached during the study period and could not be calculated.

3. Secondary Outcome: Number of Participants Who Died
Description: The number of participants who died from any cause was reported.
Time Frame: From inclusion in the study until death from any cause (maximum up to 3 years overall)
Population: ITT Population.
Measure: Number; unit: participants
Arm/Group | Erlotinib | Placebo
Number analyzed (Participants) | 46 | 48
participants | 7 | 5

4. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from inclusion in the study to date of death for any reason. The median duration of OS and corresponding 95% CI were to be estimated by Kaplan-Meier analysis and expressed in months.
Time Frame: From inclusion in the study until death from any cause (maximum up to 3 years overall)
Population: ITT Population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Erlotinib | Placebo
Number analyzed (Participants) | 46 | 48
months | NA [NA to NA] — The lower limit of the 95% CI for OS was not reached during the study period and therefore no values could be calculated. | NA [NA to NA] — The lower limit of the 95% CI for OS was not reached during the study period and therefore no values could be calculated.

ADVERSE EVENTS:
Time Frame: From Baseline until end of treatment (up to 1 year)
Description: ITT Population. Adverse events (AEs) are organized by Medical Dictionary for Regulatory Activities (MedDRA) System Organ Class (SOC), but the AE terms included below are same as they were originally registered and saved.
Arm/Group | Erlotinib | Placebo
Serious Adverse Events (participants affected / at risk) | 4/46 | 2/48
Other Adverse Events (participants affected / at risk) | 36/46 | 31/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib (N=46) | Placebo (N=48)
Respiratory tract infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Dental extraction (Surgical and medical procedures) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Aneurism (Vascular disorders) | 1 | 0
Resection of right cervical tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib (N=46) | Placebo (N=48)
Anemia (Blood and lymphatic system disorders) | 2 | 4
Acufenos (Ear and labyrinth disorders) | 2 | 3
Earache (Ear and labyrinth disorders) | 4 | 2
Dry mouth (Gastrointestinal disorders) | 12 | 18
Diarrhea (Gastrointestinal disorders) | 12 | 0
Dysphagia (Gastrointestinal disorders) | 6 | 7
Dyspesia (Gastrointestinal disorders) | 3 | 2
Stomatitus (Gastrointestinal disorders) | 2 | 3
Odynophagia (Gastrointestinal disorders) | 1 | 9
Asthenia (General disorders) | 15 | 11
Edema (General disorders) | 3 | 5
Localized edema (General disorders) | 4 | 4
Mucosa inflammation (General disorders) | 7 | 5
Pyrexia (General disorders) | 5 | 0
Folliculitis (Infections and infestations) | 7 | 1
Anorexia (Metabolism and nutrition disorders) | 5 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 5 | 5
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 | 3
Musculoskeletal rigidity (Musculoskeletal and connective tissue disorders) | 3 | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 5
Acne (Skin and subcutaneous tissue disorders) | 6 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 7 | 1
Rash (Skin and subcutaneous tissue disorders) | 8 | 1
Skin toxicity (Skin and subcutaneous tissue disorders) | 5 | 0

LIMITATIONS AND CAVEATS:
The Study was terminated early as a result of slow recruitment. Results should be interpreted with consideration of the small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.